CLINICAL TRIAL: NCT05692973
Title: The Role of Knowledge Retrieval in Inference-making Among Struggling Readers
Brief Title: The Role of Knowledge Retrieval in Inference-making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Jewell College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2026_aebarth
Record Dates: First submitted 2022-11-02; First posted 2023-01-20 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Reading Disability; Reading Problem
Keywords: Inference-making; Knowledge retrieval; Reading comprehension
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: In year 1 , Participants will be randomized to a variable test condition; repeated test condition; or a placebo condition to determine if the retrieval of knowledge through testing leads to improved inference making. In year 2, participants in the variable and repeated test conditions will receive a short intervention to determine if direct instruction in inferencing leads to improved inferencing and comprehension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Variable Test (Experimental): Students will be taught a knowledge base comprised of 18 facts about Egypt. After learning the knowledge base to criterion, students will practice retrieving the knowledge base across four testing sessions spaced 24 hours apart. Students will receive different questions across testing sessions. Next, students will read 6 passages about Egypt and then answer literal and inferential questions about the passages. Immediately after reading the passages, students will get re-tested on their retention of the knowledge base and use of the knowledge base to form inferences. They will also get retested one week and one month later to examine students' long-term retention of the knowledge base and use to make inferences.
  Interventions: Behavioral: Role of Knowledge Retrieval; Behavioral: Inference Intervention
- Repeated Test (Experimental): Students will be taught a knowledge base comprised of 18 facts about Egypt. After learning the knowledge base to criterion, students will practice retrieving the knowledge base across four testing sessions spaced 24 hours apart. Students will receive the same questions repeated across testing sessions. Next, students will read 6 passages about Egypt and then answer literal and inferential questions about the passages. Immediately after reading the passages, students will get re-tested on their retention of the knowledge base and use of the knowledge base to form inferences. They will also get retested one week and one month later to examine students' long-term retention of the knowledge base and use to make inferences.
  Interventions: Behavioral: Role of Knowledge Retrieval; Behavioral: Inference Intervention
- Placebo (Placebo Comparator): Students will be taught a knowledge base comprised of 18 facts about Egypt. After learning the knowledge base to criterion, students will re-read the passages. They will not receive any questions. Next, students will read 6 passages about Egypt and then answer literal and inferential questions about the passages. Immediately after reading the passages, students will get re-tested on their retention of the knowledge base and use of the knowledge base to form inferences. They will also get retested one week and one month later to examine students' long-term retention of the knowledge base and use to make inferences.
  Interventions: Behavioral: Role of Knowledge Retrieval; Behavioral: Inference Intervention

INTERVENTIONS:
Behavioral: Role of Knowledge Retrieval — Students will learn a new knowledge base to perfect mastery. Following the attainment of mastery students will read passages on the topic and answer questions that prompt the literal recall of key facts and the formation of inferences.
Behavioral: Inference Intervention — The intervention will pre-teach students a set of 20 essential facts about Egypt. Students will interact with expository and narrative texts. Students will practice using a text clue strategy to activate and integrate prior knowledge, will make in-text connections, connections across the 3 intervention texts, and connections between text and knowledge, and will make inferences about character motives and author intent. The tutor will ask students to justify connections and evaluate how these connections enhance understanding. Students will answer inference questions that require using text and background knowledge. A simple graphic organizer will support and scaffold inferencing. Throughout the intervention, students will practice retrieving the 20 essential facts about Egypt from memory using flash cards, completed in pairs with students providing each other feedback.

SUMMARY:
This project will (a) examine the relationship between knowledge retrieval and inferencing; (b) determine the effectiveness of an intervention that improves knowledge retrieval and inferencing among struggling readers; and (c) expand research opportunities for undergraduates. The research design uses 316 struggling readers in grades 4-6 of diverse backgrounds. The effects of knowledge retrieval (accuracy and speed) on inferencing will be modeled without dichotomizing the distribution. Linear mixed effect models will be fit to determine whether reader characteristics make unique contributions to inferencing across the posttest and follow-up data collection time points. First, several structural models will be considered as students may be nested in teachers, schools, and tutors. Unconditional models will estimate the intraclass correlation for each level of the study design. If significant interclass correlations emerge, multilevel models will be fit to evaluate the effectiveness of the intervention while controlling for covariates such as pre-test performance on inference-related measures and child-attributes such as English learner status. The primary analysis plan assumes an intent-to-treat model in which the efficacy of two intact conditions will be tested. Effect sizes will be estimated to report the magnitude of difference between the two conditions. Expected outcomes include (a) the identification of a method that effectively facilitates knowledge retrieval and the application of relevant knowledge to form inferences among elementary struggling readers from diverse backgrounds; (b) the validation of an intervention that teaches struggling readers how to activate, retrieve, and interweave relevant knowledge with information in the text and accurately form inferences while reading that can be broadly implemented in general education classrooms; and (c) expansion of undergraduate research opportunities, particularly among students from diverse backgrounds who have been historically underserved.

DETAILED DESCRIPTION:
Theory and research suggest that inferencing serves as a critical aspect of comprehension and that inferencing fails when readers do not possess sufficient background knowledge or slowly retrieve and integrate knowledge from memory or text when reading. Research suggests that readers fluently retrieve and use knowledge that is well-connected to form inferences while reading. Further, inferencing among skilled comprehenders depends considerably on knowledge retrieval, thus implicating the important role knowledge plays in inferencing. Yet, very little research has examined how inferencing changes as a function of changes in knowledge. Understanding how inferencing adapts as a function of knowledge acquisition and knowledge use provides a necessary mechanism for refining how to improve this learning process, especially for older students with reading comprehension difficulties. This project fills this critical need. This project's goal is to determine if knowledge retrieval is a mechanism for improving inferencing among middle grade struggling readers attending rural schools. The central hypothesis is that knowledge is malleable, with fluent retrieval of relevant knowledge associated with improved inferencing. This hypothesis will be tested with the objective to evaluate knowledge retrieval methods and then test the effectiveness of an intervention that facilitates knowledge retrieval and inferencing among middle grade struggling readers attending rural schools. This proposal is scientifically important because it informs theory by determining whether fluent retrieval of relevant knowledge enables inferencing among struggling readers. It is practically important because it identifies the learning strategies struggling readers need to retrieve knowledge to make inferences. The rural context also becomes critically important here. Long-standing disparities in educational access exist for students of minority backgrounds, English-learners, and children at risk for learning disabilities who attend rural schools. However, fully powered randomized control trials rarely occur in rural settings and existing literature of studies in rural schools commonly contains methodological limitations. These gaps in the literature will be addressed through the following Aims.

Aim 1: Evaluate the relationship between knowledge retrieval and inferencing. This Aim will examine whether retrieval practice - a powerful and proven technique for enhancing knowledge retrieval, inferencing, and transfer among skilled adult readers - also improves knowledge retrieval and inferencing among rural, middle grade, struggling readers. Past research conducted in the middle grades shows that retrieval practice is associated with improved end-of-unit performance in content area classrooms. But no study has examined how, why, when, and for whom knowledge retrieval works and under what conditions for struggling readers. The primary hypothesis is that fluent retrieval of relevant knowledge facilitates inferencing. The expected outcome is the identification of a method that effectively facilitates knowledge retrieval and the application of relevant knowledge to form inferences among rural, middle grade, struggling readers.

Aim 2: Determine the effectiveness of an intervention that improves knowledge retrieval and inferencing. No intervention study has used knowledge retrieval techniques to help struggling readers retain new knowledge or retrieve and use relevant knowledge to form inferences while reading. The primary hypothesis is that changes in inferencing are associated with changes in knowledge retrieval; however, knowledge retrieval and inferencing must be explicitly taught and sufficiently practiced for inferencing to occur with the same regularity as skilled comprehenders use it. The expected outcome is the validation of an intervention that teaches rural, struggling middle grade readers how to activate, retrieve, and interweave relevant knowledge with information in the text to accurately form inferences while reading. Furthermore, very few reading intervention studies have occurred with middle grade struggling readers attending rural schools. The rural setting is important; existing practices do not consider the cumulative effects of rural poverty on general knowledge development and reading achievement or the long-term impact of limited access to academic support services. Additionally, only one inference intervention study has included English Learners. The English Learner population has increased substantially in rural communities, but past research shows that generalizing vocabulary and knowledge building interventions designed for monolinguals have not proven effective.

Aim 3. To expand undergraduate research opportunities by integrating undergraduate students on the research team with the knowledge and skills to successfully implement these randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* performance below a a standard score of 93 on the Test of Silent Reading Efficiency

Exclusion Criteria:

* clinical diagnosis of a significant cognitive impairment
* clinical diagnosis of a significant behavioral disability

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gates-MacGinite Reading Test-4th Edition; Change is being assessed | pre-intervention
  a standardized, group-administered, multiple-choice assessment of reading comprehension.
Gates-MacGinite Reading Test-4th Edition; change is being assessed | immediately after the intervention
  a standardized, group-administered, multiple-choice assessment of reading comprehension
Test of Language Competence-Expanded; Change is being assessed | pre-intervention
  Inference Task asks students to read three sentences and form an inference
Test of Language Competence-Expanded; change is being assessed | immediately after the intervention
  Inference Task asks students to read three sentences and form an inference
Bridge-IT; change is being assessed | pre-intervention
  asks students to read a five-sentence text, form an inference, and determine if the next sentence provided continues the story.
Bridge-IT; change is being assessed | immediately after the intervention
  asks students to read a five-sentence text, form an inference, and determine if the next sentence provided continues the story.
Clinical Evaluation of Language Fundamentals-5; change is being assessed | pre-intervention
  Metalinguistics, Making Inferences subtest, an individually administered assessment, measures students' ability to make gap-filling inferences on the basis of causal relationships or event chains depicted in short narratives that are presented both orally and in print form.
Clinical Evaluation of Language Fundamentals-5; change is being assessed | immediately after the intervention
  Metalinguistics, Making Inferences subtest, an individually administered assessment, measures students' ability to make gap-filling inferences on the basis of causal relationships or event chains depicted in short narratives that are presented both orally and in print form.

SECONDARY OUTCOMES:
Knowledge Retrieval; change is being assessed | pre-intervention
  It teaches new knowledge then measures the accuracy and efficiency by which the individual can retrieve that knowledge. After learning the knowledge base, students read passages and form inferences with the accuracy and efficiency of inferencing measured.
Knowledge Retrieval; change is being assessed | Immediately after the intervention
  It teaches new knowledge then measures the accuracy and efficiency by which the individual can retrieve that knowledge. After learning the knowledge base, students read passages and form inferences with the accuracy and efficiency of inferencing measured.
Knowledge Retrieval; change is being assessed | one-week after the intervention
  It teaches new knowledge then measures the accuracy and efficiency by which the individual can retrieve that knowledge. After learning the knowledge base, students read passages and form inferences with the accuracy and efficiency of inferencing measured.
Knowledge Retrieval; change is being assessed | one-month after the intervention
  It teaches new knowledge then measures the accuracy and efficiency by which the individual can retrieve that knowledge. After learning the knowledge base, students read passages and form inferences with the accuracy and efficiency of inferencing measured.
Test of Word Reading Efficiency-2; change is being assessed | pre-intervention
  Sight Word Efficiency, a 45-second assessment of students' word reading accuracy and speed and Phonemic Decoding Efficiency, a 45-second assessment of students' non-word reading accuracy and speed.
Test of Word Reading Efficiency-2; change is being assessed | immediately after the intervention
  Sight Word Efficiency, a 45-second assessment of students' word reading accuracy and speed and Phonemic Decoding Efficiency, a 45-second assessment of students' non-word reading accuracy and speed.
Metacognition survey; change is being assessed | pre-intervention
  asks students to report study strategies used when learning from text and includes questions about repeated studying and retrieval practice.
Metacognition survey; change is being assessed | immediately after the intervention
  asks students to report study strategies used when learning from text and includes questions about repeated studying and retrieval practice.
Contextualized Reading Strategy Survey; change is being assessed | pre-intervention
  49-item self-report survey designed to assess a collection of learning and comprehension strategies that students might use when reading for school.
Contextualized Reading Strategy Survey; change is being assessed | immediately after the intervention
  49-item self-report survey designed to assess a collection of learning and comprehension strategies that students might use when reading for school.
Working Memory Test Battery for Children | pre-intervention
  Word List Recall that asks the student to repeat a list of monosyllabic words, Non-word List Recall that asks the student to repeat a list of non-words and Listening Recall Test that requires that the student listen to a series of short sentences, judge their accuracy, and recall the final word of each sentence.
Kauffman Brief Intelligence Test-2 | pre-intervention
  Verbal Knowledge subtest, a norm-referenced, individually administered assessment of expressive word and world knowledge
Gates-MacGinitie Vocabulary Test; change is being assessed | pre-intervention
  group administered test of receptive vocabulary
Gates-MacGinitie Vocabulary Test; change is being assessed | immediately after the intervention
  group administered test of receptive vocabulary
Egyptian Content Knowledge; change is being assessed | pre-intervention
  a researcher developed assessment of one's knowledge of Egypt
Egyptian Content Knowledge; change is being assessed | immediately after the intervention
  a researcher developed assessment of one's knowledge of Egypt
Test of Silent Reading Efficiency and Comprehension; change is being assessed | pre-intervention
  measure of silent reading fluency and understanding of text
Test of Silent Reading Efficiency and Comprehension; change is being assessed | immediately after the intervention
  measure of silent reading fluency and understanding of text
Test of Silent Contextual Reading Fluency; change is being assessed | pre-intervention
  measures of silent reading fluency and understanding of text
Test of Silent Contextual Reading Fluency; change is being assessed | immediately after the intervention
  measures of silent reading fluency and understanding of text
CBM-Maze Task; change is being assessed | pre-intervention
  measure of silent reading fluency and understanding of text
CBM-Maze Task; change is being assessed | immediately after the intervention
  measure of silent reading fluency and understanding of text

OTHER OUTCOMES:
Test of Silent Reading Efficiency and Comprehension | baseline screening of participants; pre-intervention
  measure of silent reading fluency and understanding of text

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Barth, Ph.D, Principal Investigator — William Jewell College
Locations (1):
- Excelsior Springs School District, Excelsior Springs, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The following steps will be enacted: (a) requester will submit an email to the PI requesting data sharing; (b) A data-sharing agreement will be forwarded to the requester by the laboratory manager; (c) once the data-Sharing agreement is returned, a file will be prepared for the requester. This file will be prepared by PI or the laboratory manager; (d) files will be shared via secure data archive. Our data archives are secure and approved for use with Category I data.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available at the close of the project.
Access Criteria: Data will be available upon request. A data-sharing agreement will be required prior to release of data. The agreement will include a summary of the purpose of the data, methodology and procedures used to the collected the data, timing of the data use. The agreement will also state that privacy and confidentiality standards will be maintained and that manipulation of data for the purposes of identifying subjects is prohibited.

REFERENCES:
- [Background] Barth AE, Elleman A. Evaluating the Impact of a Multistrategy Inference Intervention for Middle-Grade Struggling Readers. Lang Speech Hear Serv Sch. 2017 Jan 1;48(1):31-41. doi: 10.1044/2016_LSHSS-16-0041. PMID 27776201
- [Background] Barth AE, Daniel J, Roberts G, Vaughn S, Barnes MA, Ankrum E, Kincaid H. The Role of Knowledge Availability in Forming Inferences with Rural Middle Grade English Learners. Learn Individ Differ. 2021 May;88:102006. doi: 10.1016/j.lindif.2021.102006. Epub 2021 May 12. PMID 33994756

DOCUMENTS (2):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT05692973/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT05692973/SAP_001.pdf